CLINICAL TRIAL: NCT01979809
Title: Encouraging Young Adults to Make Effective Nutrition Choices: MENU GenY Study
Brief Title: Encouraging Young Adults to Make Effective Nutrition Choices
Acronym: MENU GenY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Geisinger Clinic (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Gwen Alexander, PhD, Assistant Research Scientist, Henry Ford Health System
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD067314-01A1 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Improve Dietary Behaviors in Young Adults 21-30 Years of Age
Keywords: Dietary change; Young adult; Prevention; Web-based intervention; eCoaching

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Sham Comparator): Untailored control website designed to support increase in fruit and vegetables with no age targeting used in previously funded MENU Choices study
  Interventions: Behavioral: MENU GenY
- Arm 2 (Active Comparator): MENU GenY age-targeted and tailored interactive website including 8 information sessions over 4 months, and options to visit over 185 recipes, videos, 4 bloggers, and information articles on dietary change topics
  Interventions: Behavioral: MENU GenY
- Arm 3 (Active Comparator): Web intervention that is age targeted and tailored, identical to Arm 2, with the addition of personalized "e-coaching" support via email.
  Interventions: Behavioral: MENU GenY

INTERVENTIONS:
Behavioral: MENU GenY — Participants will assess eligibility, complete consent and baseline survey to enroll online, then be randomized to one of 3 arms: Control Arm 1 - a non-tailored intervention with no age targeting; Arm 2 -age targeted, tailored website set to appeal to young adults and offer a varety of support using muli-media to improve dietary intake of fruit, vegetables and whole grains, and decrease sweet drinks. Arm 3 utilizes the same intervention as Arm 2, and has support via email from eCoaches who use a Motivational Interview approach to support to help change dietary patterns. All arms are active for 4 months with occasionalemail contact throughout the following 8 mo. Follow-up surveys occur at 3 mo, 6 mo, and primary outcome at 12 months.
  Other Names: MENU Choices; MENU Gen-Y; Making Effective Nutrition Choices for Young Adults: the MENU Gen-Y Study

SUMMARY:
The purpose of this study is to conduct a two site, three arm randomized intervention study to improve fruit and vegetable intake, improve whole grain intake and reduce sweetened beverages in young adults aged 21 to 30 years. This work is potentially very high impact in light of growing overweight and obesity and decreased health status overall, and potential dietary benefits to children of our target age group.

DETAILED DESCRIPTION:
In support of NIH goals to improve people's health and support a healthy lifestyle, we will conduct a randomized trial to evaluate an age-targeted web-based intervention designed to improve the diet of a young adults (ages 21-30) as they navigate a new life stage of greater independence. The goal of our study is to increase daily intake of fruits and vegetables(FV) for young adults born in or after 1980, known as "Generation Y" (GenY), using relevant features that appeal to this group. This five-year project has two phases. In the first phase, we will use focus groups to confirm planned, key intervention elements that target needs and preferences of GenY and will build engagement in the intervention, as we revise our tested, effective Internet- based intervention (Making Effective Nutrition Choices or MENU, U19-CA079689). The MENU study was designed to support an increase in FV intake, and relied solely on e-media (internet and email). In the proposed study we will revise the MENU curriculum, applying age-targeted and theory-based methods to improve intervention engagement and effectiveness for GenY dietary behavior change. The intervention will use three psychosocial features which have been subject to empirical examination by age group: Social Cognitive Theory, Self-Determination Theory (SDT), with special attention to Social Marketing Theory(SMT), which emphasizes understanding the total environment to better shape health communications.

In developing our program, we will apply knowledge about GenY from developmental psychology,guided by our consultants and formative research on individual, environmental and societal factors collected in our preliminary studies and Phase I GenY focus groups. Focus group members will evaluate our validated MENU intervention, as well as our revised age-targeted, interactive "MENU GenY" intervention prior to launch. In the second phase, we will evaluate the efficacy of the MENU GenY interventions, including the added value of the self-initiated, personalized e-coaching support by email, as a supplement to the tailored online intervention. Specifically, using a sample of 1624 adults,ages 21 - 30 and from two geographically distinct regions (urban Detroit and rural Pennsylvania), and employing a randomized, three arm design, the primary aims of Phase II are to 1) determine if an agetargeted,tailored web-based intervention is more efficacious in improving primary outcome of daily intake of FV compared to an untailored intervention arm with no age targeting (control arm); 2) determine if a tailored webbased intervention with age targeting and personalized e-coaching support is more efficacious than the control; and 3) determine if the tailored web-based intervention with age targeting and e-counseling is more efficacious than a tailored web-based intervention with age targeting alone.

ELIGIBILITY:
Inclusion Criteria:

* 21-30 years of age
* receive medical care from Henry Ford Health System (Detroit, MI) or Geisinger Health System (Danville area and central Pennsylvania)

Exclusion Criteria:

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1674 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

PRIMARY OUTCOMES:
Change in fruit and vegetable intake at 12 months post enrollment, 2-item screener and CDC 24 hour screener | Primary assessm't is 12 months post enrollment
  Using the 2-item fruit and vegetable screener and CDC screener, which will be used to assess fruit and vegetable intake at baseline, 3 months, 6 months and 12 months. Also, to be examined is variation in dietary change by contextual factors including site, demographics, program engagement, environment, social and motivational factors.

SECONDARY OUTCOMES:
CDC screener to measure sweetened beverage intake | 12 months
  Compare baseline intake of sweetened beverages to assessments at 3 month, 6 month and 12 months post enrollment.
CDC screener to measure increase in whole grains | 12 months
  Utilizling the CDC food screener, we will assess change in whole grain consumption at baseline and compare findings at 3 months, 6 months, and 12 monthspost enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Alexander, Ph.D, Principal Investigator — Henry Ford Health System
Locations (2):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - Geisinger Health System, Danville, Pennsylvania